CLINICAL TRIAL: NCT01223105
Title: Longitudinal Evaluation of Vitrification of Human Oocytes
Brief Title: Oocyte Cryopreservation by Slow Freezing and Vitrification
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMA-2009-02
Record Dates: First submitted 2010-10-08; First posted 2010-10-18 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Women Diagnosed With Cancer; Egg Donors; Single Women; Failed Sperm Procurement in IVF
Keywords: slow freeze; cryopreservation; vitrification; oocyte preservation
MeSH Terms: interventions — Cryopreservation; Vitrification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Slow Freezing (Experimental): oocytes will be frozen by slow freeze/ rapid thaw
  Interventions: Procedure: slow freeze
- Vitrification (Experimental): oocytes will be frozen using rapid freezing/rapid thaw
  Interventions: Procedure: Vitrification

INTERVENTIONS:
Procedure: slow freeze — Eggs will be placed in a cryo-protected solution and frozen slowly in a programable freezer
  Other Names: Cryopreservation; Traditional freezing; slow freezing
  Arms: Slow Freezing
Procedure: Vitrification — Eggs will be placed in a high concentration of cryo-protectant and frozen very quickly by plunging in liquid nitrogen
  Arms: Vitrification

SUMMARY:
This study seeks to evaluate whether the vitrification technique, as compared to the more traditional slow-cooling technique, leads to higher rates of successful thawing, fertilization, implantation and delivery.

DETAILED DESCRIPTION:
Cryopreservation (freezing) of human gametes (unfertilized egg) provides a great potential to preserve or extend fertility in the face of disease and social circumstances (cancer diagnosis, delaying childbirth, single women, etc.). There are two methods for storage of oocytes (unfertilized eggs): slow freezing or vitrification (uses higher concentrations of cryoprotectant and faster cooling rates). Slow freezing is the standard method and has been successful for embryos since 1983 and more recently for oocytes. Recent reports indicate that vitrification may be more successful than slow freezing. The aim of this study is to examine the rate at which frozen eggs survive freezing and thawing, the rate at which the frozen/thawed eggs fertilize with sperm and the pregnancy outcomes of oocyte (egg) vitrification cycles to determine whether the outcomes are similar or better than standard oocyte (egg) cryopreservation (freezing) cycles.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 50 years, at the time of informed consent.
* Subjects must agree to undergo intracytoplasmic sperm injection (ICSI)

Exclusion Criteria:

* Presence of any medical condition that contraindicates ovarian stimulation, in vitro fertilization or pregnancy.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Oocytes survival after thaw | 1 month
  Whether each oocyte survives the thawing process

SECONDARY OUTCOMES:
Fertilization | 1 month
  Whether each oocyte is successfully fertilized
Implantation | 1 month
  Whether pregnancy occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, HCLD, Study Director — RMA of NJ; Kathleen Ferry, BS, Study Chair — RMA of NJ